CLINICAL TRIAL: NCT01552915
Title: A Phase 4, Randomized, Double-blind, Multicenter, Parallel-group, Active-controlled, Dose-optimization Safety and Efficacy Study of SPD489 (VYVANSE®) Compared With OROS-MPH (CONCERTA®) With a Placebo Reference Arm, in Adolescents Aged 13-17 Years With Attention-deficit/Hyperactivity Disorder (ADHD)
Brief Title: Effectiveness of Vyvanse Compared to Concerta in Adolescents With Attention-deficit/Hyperactivity Disorder
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SPD489-405
Record Dates: First submitted 2012-03-06; First posted 2012-03-13 (Estimated); Results first posted 2014-12-11 (Estimated); Last update posted 2021-06-08 (Actual); Status verified 2021-05

CONDITIONS: Attention-deficit/Hyperactivity Disorder
Keywords: ADHD
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Lisdexamfetamine Dimesylate; Methylphenidate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Lisdexamfetamine Dimesylate (Experimental)
  Interventions: Drug: Lisdexamfetamine dimesylate
- Methylphenidate Hydrochloride (Active Comparator)
  Interventions: Drug: Methylphenidate Hydrochloride
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Lisdexamfetamine dimesylate — Daily oral dosing in the AM of optimized dose, ranging from 30- 70 mg. 5 week dose optimization, 3 week dose maintenance
  Other Names: LDX, Vyvanse, SPD489
  Arms: Lisdexamfetamine Dimesylate
Drug: Methylphenidate Hydrochloride — Daily oral dosing in the AM of optimized dose, ranging from 18-72 mg. 5 week dose optimization, 3 week dose maintenance
  Other Names: OROS-MPH, Concerta
  Arms: Methylphenidate Hydrochloride
Drug: Placebo — Daily oral dosing in the AM for 8 weeks
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine effectiveness of Vyvanse compared to Concerta in adolescents with Attention-deficit/Hyperactivity Disorder (ADHD).

ELIGIBILITY:
Inclusion Criteria:

* Subject must be 13-17 years of age, inclusive, at the time of consent.
* Subject must weigh more than 79.5lb.
* The parent/LAR must be available at approximately 7:00AM (±2 hours) to dispense the dose of investigational product for the study duration.
* Subject, who is a female, must have a negative serum beta human chorionic gonadotropin (β-HCG) pregnancy test and a negative urine pregnancy test and agree to comply with any applicable contraceptive requirements of the protocol.
* Subject has an ADHD-RS-IV total score ≥28.
* Subject is able to swallow a capsule.
* Subject does not have hypertension and has a resting sitting blood pressure less than or equal to 135/85mmHg.

Exclusion Criteria

* Subject has a current, controlled (with medications prohibited in this study) or uncontrolled, comorbid psychiatric diagnosis with significant symptoms such as any significant comorbid Axis II disorder or significant Axis I disorder (such as post traumatic stress disorder, psychosis, bipolar illness, pervasive developmental disorder, severe obsessive compulsive disorder, depressive or anxiety disorder.
* Diagnosis of conduct disorder. Oppositional defiant disorder is not exclusionary.
* Subject is considered a suicide risk, has previously made a suicide attempt, or is currently demonstrating active suicidal ideation. Subjects with intermittent passive suicidal ideation are not necessarily excluded.
* Subject is underweight or overweight.
* Subject has a concurrent chronic or acute illness (such as severe allergic rhinitis or an infectious process requiring antibiotics), disability, or other condition. Mild, stable asthma is not exclusionary.
* Subject has a history of seizures (other than infantile febrile seizures), a chronic or current tic disorder, or a current diagnosis and/or a known family history of Tourette's Disorder.
* Subject has a known history of symptomatic cardiovascular disease, advanced arteriosclerosis, structural cardiac abnormality, cardiomyopathy, serious heart rhythm abnormalities, coronary artery disease, or other serious cardiac problems that may place him/her at increased vulnerability to the sympathomimetic effects of a stimulant medication.
* Subject has a known family history of sudden cardiac death or ventricular arrhythmia.
* Subject has any clinically significant ECG or clinically significant laboratory abnormality.
* Subject has current abnormal thyroid function, defined as abnormal thyroid stimulating hormone (TSH) and thyroxine (T4). Treatment with a stable dose of thyroid medication for at least 3 months is permitted.
* Subject has a documented allergy, hypersensitivity, or intolerance to amphetamine or to any excipients in the investigational product.
* Subject has a documented allergy, hypersensitivity, or intolerance to MPH or to any excipients in the reference product.
* Subject has failed to fully respond to an adequate course(s) (dose and duration) of MPH or amphetamine therapy.
* Subject has a history of suspected substance abuse or dependence disorder (excluding nicotine). Subjects with a lifetime history of amphetamine, cocaine, or other stimulant abuse and/or dependence will be excluded.
* Subject has a positive urine drug result.
* Subject has previously participated in this study or another clinical study involving SPD489/NRP104.
* Subject has glaucoma.
* Subject is required to take or anticipates the need to take medications that have CNS effects or affect performance, such as sedating antihistamines and decongestant sympathomimetics, or are monoamine oxidase inhibitors. Stable use of bronchodilator inhalers is not exclusionary.
* Subject is female and is pregnant or lactating.
* Subject is well controlled on his/her current ADHD medication.
* Subject has a pre-existing severe gastrointestinal tract narrowing.

Ages: 13 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 464 (Actual)
Dates: Start 2012-04-17 (Actual); Primary Completion 2014-01-22 (Actual); Study Completion 2014-01-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (79):
- United States (79):
  - Melmed Center, Scottsdale, Arizona
  - Clinical Study Centers, LLC, Little Rock, Arkansas
  - Synergy Clinical Research Center, National City, California
  - Pacific Clinical Research Medical Group, Orange, California
  - SDS Clinical Trials, Inc., Orange, California
  - Peninsula Research Associates, Inc., Rolling Hills Estates, California
  - PCSD - Feighner Research, San Diego, California
  - University of California, San Francisco, San Francisco, California
  - Neuropsychiatric Research Center of Orange County, Santa Ana, California
  - Elite Clinical Trials, Wildomar, California
  - MCB Clinical Research Centers, LLC, Colorado Springs, Colorado
  - Florida Clinical Research Center, LLC, Bradenton, Florida
  - Sarkis Clinical Trials, Gainesville, Florida
  - Amedica Research Institute, Hialeah, Florida
  - Clinical Neuroscience Solutions, Inc., Jacksonville, Florida
  - Fidelity Clinical Research, Inc., Lauderhill, Florida
  - Florida Clinical Research Center, LLC, Maitland, Florida
  - Scientific Clinical Research, Inc., Miami, Florida
  - Clinical Neuroscience Solutions, Inc., Orlando, Florida
  - Compass Research, LLC, Orlando, Florida
  - Stedman Clinical Trials, Tampa, Florida
  - Janus Center for Psychiatric Research, West Palm Beach, Florida
  - Atlanta Institute of Medicine and Research, Atlanta, Georgia
  - Capstone Clinical Research, Libertyville, Illinois
  - AMR Baber Research Group, Inc., Naperville, Illinois
  - AMR Conventions Research, Naperville, Illinois
  - American Medical Research, Inc, Oak Brook, Illinois
  - Advocate Hope Children's Hospital, Oak Lawn, Illinois
  - Neuroscience Research Institute, Inc, Oak Park, Illinois
  - Psychiatric Associates, Overland Park, Kansas
  - University of Kentucky, Lexington, Kentucky
  - Four Rivers Clinical Research, Paducah, Kentucky
  - Neuroscientific InSights, Rockville, Maryland
  - Marc Hertzman MD, PC, Rockville, Maryland
  - Rochester Center for Behavioral Medicine, Rochester Hills, Michigan
  - Clinical Neurophysiology Services, PC, Sterling Heights, Michigan
  - Behavioral Medical Center - Troy, Troy, Michigan
  - Precise Research Centers, Flowood, Mississippi
  - Comprehensive Psychiatric Associates, Gladstone, Missouri
  - St Charles Psychiatric Associates, Saint Charles, Missouri
  - Premier Psychiatric Research Institute, Lincoln, Nebraska
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Center for Psychiatry and Behavioral Medicine, Inc., Las Vegas, Nevada
  - Center for Emotional Fitness, Cherry Hill, New Jersey
  - CRCNJ - Clinical Research Center of New Jersey, Gibbsboro, New Jersey
  - Neurcognitive Institute, Mount Arlington, New Jersey
  - Mount Sinai School of Medicine, New York, New York
  - Duke Child and Family Study Center, Durham, North Carolina
  - Innovis Health, LLC, Fargo, North Dakota
  - North Coast Clinical Trials, Beachwood, Ohio
  - University of Cincinnati Dept. of Psychiatry & Behavioral, Cincinnati, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - The Ohio State University Nisonger Center, Columbus, Ohio
  - Midwest Clinical Research Center, Dayton, Ohio
  - Professional Psychiatric Services, Mason, Ohio
  - Family Practice of Wadsworth, Inc., Wadsworth, Ohio
  - Cyn3rgy Research, Gresham, Oregon
  - Oregon Center for Clinical Investigations, Inc. (OCCI, Inc.), Portland, Oregon
  - Summit Research Network (Oregon) Inc., Portland, Oregon
  - Oregon Center for Clinical Investigations, Inc., Salem, Oregon
  - Carolina Clinical Trials, Inc., Charleston, South Carolina
  - Coastal Carolina Research Center, Mt. Pleasant, South Carolina
  - Research Strategies of Memphis, LLC, Memphis, Tennessee
  - FutureSearch Trials, Austin, Texas
  - Claghorn-Lesem Reseach Clinic, Ltd., Houston, Texas
  - Texas Center for Drug Development, Inc., Houston, Texas
  - Red Oak Psychiatry Associates, PA, Houston, Texas
  - R/D Clinical Research, Inc., Lake Jackson, Texas
  - Westex Clinical Investigations, Lubbock, Texas
  - Clinical Trials of Texas, Inc., San Antonio, Texas
  - University of Texas HSC at San Antonio Dept. of Psychiatry, San Antonio, Texas
  - Wharton Research Center, Inc., Wharton, Texas
  - Psychiatric & Behavioral Solutions, Salt Lake City, Utah
  - University of Virginia Child and Family Psychiatry Clinical, Charlottesville, Virginia
  - NeuroScience, Inc., Herndon, Virginia
  - Northwest Clinical Research Center, Bellevue, Washington
  - Eastside Therapeutic Resource, Kirkland, Washington
  - Summit Research Network (Seattle), LLC, Seattle, Washington
  - Rockwood Clinic, P.S., Spokane, Washington

REFERENCES:
- [Derived] Newcorn JH, Nagy P, Childress AC, Frick G, Yan B, Pliszka S. Randomized, Double-Blind, Placebo-Controlled Acute Comparator Trials of Lisdexamfetamine and Extended-Release Methylphenidate in Adolescents With Attention-Deficit/Hyperactivity Disorder. CNS Drugs. 2017 Nov;31(11):999-1014. doi: 10.1007/s40263-017-0468-2. PMID 28980198

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Subjects received over encapsulated placebo that matched the SPD489 and OROS-MPH capsules.
- SPD489: Subjects received over encapsulated SPD489 titrated to an optimal dose of 30, 50, or 70mg/day
- OROS-MPH: Subjects received over encapsulated OROS-MPH titrated to an optimal dose of 18, 36, 54, or 72mg/day. Subjects optimized to 72mg received two 36mg tablets.
Period: Overall Study
Arm/Group | Placebo | SPD489 | OROS-MPH
Started | 91 (This population is from the Safety Set. Two randomized subjects were not dosed and were excluded.) | 184 (This population is from the Safety Set. Two randomized subjects were not dosed and were excluded.) | 184 (This population is from the Safety Set. One randomized subject was not dosed and was excluded.)
Completed | 68 | 155 | 157
Not Completed | 23 | 29 | 27
Not completed — Adverse Event | 3 | 14 | 3
Not completed — Lost to Follow-up | 4 | 6 | 5
Not completed — Withdrawal by Subject | 6 | 4 | 5
Not completed — Protocol Violation | 0 | 4 | 4
Not completed — Lack of Efficacy | 8 | 1 | 4
Not completed — Other | 2 | 0 | 6

BASELINE CHARACTERISTICS:
Population: Safety Set: All subjects in the Randomized Set who took at least 1 dose of investigational product.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | SPD489 | OROS-MPH | Total
Number analyzed (Participants) | 91 | 184 | 184 | 459
Age, Continuous [Mean (Standard Deviation); unit: Years] | 14.8 (1.43) | 14.7 (1.38) | 14.7 (1.32) | 14.7 (1.37)
Age, Customized [Count of Participants; unit: Participants]
  <=18 years | 91 | 184 | 184 | 459
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30 | 62 | 62 | 154
  Male | 61 | 122 | 122 | 305
Region of Enrollment [Count of Participants; unit: Participants]
  UNITED STATES | 91 | 184 | 184 | 459

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Attention-Deficit/Hyperactivity Disorder Rating Scale, Fourth Edition (ADHD-RS-IV) Total Score at Week 8
Description: The ADHD-RS-IV consists of 18 items scored on a 4-point scale ranging from 0 (no symptoms) to 3 (severe symptoms) with total score ranging from 0 to 54. Higher score indicates more severe symptoms.
Time Frame: Baseline and week 8
Population: Full Analysis Set: All subjects who took at least 1 dose of investigational product and who had at least 1 post-baseline primary efficacy assessment.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | SPD489 | OROS-MPH
Number analyzed (Participants) | 89 | 179 | 184
units on a scale | -13.4 (1.19) | -25.6 (0.82) | -23.5 (0.80)
Statistical Analysis 1: Comparison: SPD489 vs OROS-MPH; Test type: Superiority or Other; p = 0.0717, mixed effects model for repeated measure; Difference in LS Mean = -2.1, 95% CI 2-sided [-4.3 to 0.2], Standard Error of Mean 1.15
Statistical Analysis 2: Comparison: Placebo vs SPD489; Test type: Superiority or Other; p < 0.0001, mixed effects model for repeated measure; Difference in LS Mean = -12.2, 95% CI 2-sided [-15.1 to -9.4], Standard Error of Mean 1.45
Statistical Analysis 3: Comparison: Placebo vs OROS-MPH; Test type: Superiority or Other; p < 0.0001, mixed effects model for repeated measure; Difference in LS Mean = -10.1, 95% CI 2-sided [-13.0 to -7.3], Standard Error of Mean 1.43

2. Secondary Outcome: Percentage of Participants With Improvement on Clinical Global Impression - Global Improvement (CGI-I) at Week 8 - Last Observation Carried Forward (LOCF)
Description: Clinical Global Impression-Improvement (CGI-I) consists of a 7-point scale ranging from 1 (very much improved) to 7 (very much worse). Improvement is defined as a score of 1 (very much improved) or 2 (much improved) on the scale.
Time Frame: Week 8
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | SPD489 | OROS-MPH
Number analyzed (Participants) | 89 | 178 | 184
percentage of participants | 34.8 | 83.1 | 81.0
Statistical Analysis 1: Comparison: SPD489 vs OROS-MPH; Test type: Superiority or Other; p = 0.6165, Cochran-Mantel-Haenszel
Statistical Analysis 2: Comparison: Placebo vs SPD489; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel
Statistical Analysis 3: Comparison: Placebo vs OROS-MPH; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel

3. Secondary Outcome: Change From Baseline in Systolic Blood Pressure at up to 8 Weeks - Last on Treatment Assessment
Time Frame: Baseline and up to 8 Weeks
Population: Safety Set: All randomized subjects who took at least 1 dose of investigational product.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Placebo | SPD489 | OROS-MPH
Number analyzed (Participants) | 89 | 179 | 184
mmHg | -0.8 (8.97) | 2.4 (9.46) | 0.4 (9.90)

4. Secondary Outcome: Change From Baseline in Diastolic Blood Pressure at up to 8 Weeks - Last on Treatment Assessment
Time Frame: Baseline and up to 8 weeks
Population: Safety Set: All randomized subjects who took at least 1 dose of investigational product.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Placebo | SPD489 | OROS-MPH
Number analyzed (Participants) | 89 | 179 | 184
mmHg | -1.2 (8.11) | 2.8 (8.41) | 2.2 (8.64)

5. Secondary Outcome: Change From Baseline in Pulse Rate at up to 8 Weeks - Last on Treatment Assessment
Time Frame: Baseline and up to 8 weeks
Population: Safety Set: All randomized subjects who took at least 1 dose of investigational product.
Measure: Mean (Standard Deviation); unit: bpm
Arm/Group | Placebo | SPD489 | OROS-MPH
Number analyzed (Participants) | 89 | 179 | 184
bpm | 0.3 (11.32) | 4.7 (11.82) | 6.0 (10.52)

ADVERSE EVENTS:
Time Frame: Duration of the study, for up to 8 weeks per participant
Description: Treatment-Emergent Adverse Events
Groups:
- SPD489: Subjects received over encapsulated SPD489 optimized among a 30, 50, or 70mg dose.
- OROS-MPH: Subjects received over encapsulated OROS-MPH optimized among a 18, 36, 54 or 72mg dose. Subjects optimized to 72mg received two 36mg tablets.
Arm/Group | Placebo | SPD489 | OROS-MPH
Serious Adverse Events (participants affected / at risk) | 0/91 | 1/184 | 1/184
Other Adverse Events (participants affected / at risk) | 39/91 | 139/184 | 120/184
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=91) | SPD489 (N=184) | OROS-MPH (N=184)
Suicidal ideation (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Renal cyst (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=91) | SPD489 (N=184) | OROS-MPH (N=184)
Abdominal pain upper (Gastrointestinal disorders) | 4 (6) | 12 (12) | 10 (13)
Dry mouth (Gastrointestinal disorders) | 1 (1) | 15 (17) | 11 (11)
Nausea (Gastrointestinal disorders) | 4 (4) | 14 (14) | 15 (17)
Fatigue (General disorders) | 3 (3) | 10 (10) | 5 (5)
Irritability (General disorders) | 9 (9) | 37 (41) | 14 (17)
Nasopharyngitis (Infections and infestations) | 1 (1) | 11 (12) | 13 (13)
Upper respiratory tract infection (Infections and infestations) | 8 (9) | 9 (9) | 6 (6)
Heart rate increased (Investigations) | 0 (0) | 8 (8) | 11 (12)
Weight decreased (Investigations) | 1 (1) | 37 (43) | 24 (26)
Decreased appetite (Metabolism and nutrition disorders) | 7 (8) | 98 (118) | 77 (85)
Dizziness (Nervous system disorders) | 1 (1) | 12 (13) | 8 (9)
Headache (Nervous system disorders) | 7 (8) | 28 (38) | 28 (35)
Somnolence (Nervous system disorders) | 4 (5) | 10 (10) | 6 (6)
Initial insomnia (Psychiatric disorders) | 2 (2) | 15 (17) | 12 (16)
Insomnia (Psychiatric disorders) | 0 (0) | 16 (17) | 15 (15)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If a multicenter publication is not submitted within twelve (12) months after conclusion, abandonment or termination of the Study at all sites, or after Sponsor confirms there shall be no multicenter Study publication, the Institution and/or such Principal Investigator may publish the results from the Institution site individually.